CLINICAL TRIAL: NCT04463719
Title: Adequate Selection of Patients for Thyroid Biopsy: Evaluation of a Shared Decision Making Conversation Aid
Brief Title: AIM2: Adequate Selection of Patients for Thyroid Biopsy: Evaluation of a Shared Decision Making Conversation Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202000837-N; 1K08CA248972-01 (NIH); 5K08CA248972-02 (NIH); OCR34613 (Other: UF OnCore)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Nodules; Thyroid Cancer
Keywords: thyroid nodules; shared decision making
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Counseling using the electronic conversation aid
  Interventions: Behavioral: Counseling using the electronic conversation aid
- Control Group (Active Comparator): Routine counseling only
  Interventions: Behavioral: counseling by routine care

INTERVENTIONS:
Behavioral: Counseling using the electronic conversation aid — Patients receive counseling about thyroid biopsy with the use of the conversation aid.
  Arms: Intervention group
Behavioral: counseling by routine care — Patients receive counseling by routine care without the use of the conversation aid
  Arms: Control Group

SUMMARY:
There is an epidemic of thyroid cancer that is harmful to patients and the medical system. The study hypothesizes that the use of an electronic conversation aid during clinical visits can help patients and clinicians collaborate. The study aims to update a conversation aid prototype that was developed to support shared decision making in the diagnosis of thyroid cancer and conduct a pilot clinical trial to evaluate the feasibility of conducting a larger efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old presenting for evaluation of a thyroid nodule

Exclusion Criteria:

* Patients with hyperthyroidism
* Patients with previous biopsy of the nodule of interest
* Pregnant patients
* Prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naykky Singh Ospina, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Intervention Group: Counseling using the electronic conversation aid
  Counseling using the electronic conversation aid: Patients receive counseling about thyroid biopsy with the use of the conversation aid.
- Patient Control Group: Routine counseling only
  counseling by routine care: Patients receive counseling by routine care without the use of the conversation aid
- Clinicians: Clinicians enrolled in the study counseled patients with or without the use of the conversation aid, per patient randomization assigment
Period: Overall Study
Arm/Group | Patient Intervention Group | Patient Control Group | Clinicians
Started | 45 | 45 | 17
Completed | 43 | 43 | 17
Not Completed | 2 | 2 | 0
Not completed — Exclusion criteria identified during clinical visit | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Information collected on the 43 patients in each group who were eligible for the study. No additional information was collected for clinicians.
Groups:
- Patients - Intervention Group: Counseling using the electronic conversation aid
  Counseling using the electronic conversation aid: Patients receive counseling about thyroid biopsy with the use of the conversation aid.
- Patients - Control Group: Routine counseling only
  counseling by routine care: Patients receive counseling by routine care without the use of the conversation aid
- Clinicians: Clinicians enrolled in the study counseled patients with or without the use of the conversation aid, per patient randomization assignment
- Total: Total of all reporting groups
Arm/Group | Patients - Intervention Group | Patients - Control Group | Clinicians | Total
Number analyzed (Participants) | 43 | 43 | 17 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No additional information was collected for clinicians.
  years
    number analyzed (Participants) | 43 | 43 | 0 | 86
    (all) | 57.1 (16.2) | 57.2 (15.5) |  | 57.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No additional information was collected on clinicians
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    Female | 36 | 33 |  | 69
    Male | 7 | 10 |  | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: No additional information was collected for clinicians
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    Hispanic or Latino | 2 | 0 |  | 2
    Not Hispanic or Latino | 41 | 43 |  | 84
    Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: No additional information was collected for clinicians.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    American Indian or Alaska Native | 0 | 1 |  | 1
    Asian | 2 | 0 |  | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Black or African American | 2 | 5 |  | 7
    White | 37 | 37 |  | 74
    More than one race | 1 | 0 |  | 1
    Unknown or Not Reported | 1 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 17 | 86
General Health [Count of Participants; unit: Participants] — Population: No additional information was collected for clinicians.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    Excellent/Very good | 20 | 10 |  | 30
    Fair | 5 | 9 |  | 14
    Good | 15 | 21 |  | 36
    Poor | 3 | 1 |  | 4
    Missing | 0 | 2 |  | 2
Education [Count of Participants; unit: Participants] — Population: No additional information was collected for clinicians.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    High school graduate | 4 | 4 |  | 8
    Graduate or professional degree | 22 | 19 |  | 41
    Less than high school | 1 | 0 |  | 1
    Professional degree in health related sciences | 5 | 6 |  | 11
    Some college, no degree | 10 | 11 |  | 21
    Missing | 1 | 3 |  | 4
Income [Count of Participants; unit: Participants] — Population: No additional information was collected for clinicians.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    >$150,000 | 7 | 6 |  | 13
    $40,000 to $79,999 | 9 | 10 |  | 19
    $80,000 to $149,999 | 11 | 11 |  | 22
    < $40,000 | 14 | 13 |  | 27
    Missing | 2 | 3 |  | 5
Thyroid nodule size [Median (Inter-Quartile Range); unit: cm] — Population: No additional information was collected for clinicians, also variable not applicable to clincians
  cm
    number analyzed (Participants) | 43 | 43 | 0 | 86
    (all) | 1.6 [1.2 to 2.6] | 1.8 [1.2 to 2.6] |  | 1.7 [1.2 to 2.6]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Patients for Feasibility
Description: Proportion of participants that are eligible relative to total trial referrals.To measure the proportion of eligible patients after review of upcoming clinical visits, enrollment and refusal reasons, ability to randomize patients and tolerability by patients and clinicians of the required assessments (time to complete assessments and obtain complete assessment at 6 months of follow up).
Time Frame: at 6 months of follow up
Population: Number of patients that were screened for inclusion in the study
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patient for the Study: Eligible patients for the study and for randomization
Arm/Group | Eligible Patient for the Study
Number analyzed (Participants) | 531
Participants
  Eligible Patients Based on Chart Review | 213
  Patients not eligible based on chart review | 318

2. Secondary Outcome: Patient's Acceptance to Participate in the Study
Description: From eligible patients that were invited to participate, the proportion of patients that agreed to enter the study
Time Frame: first visit
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients Invited to Participate in the Study: All patients that were eligible and invited to participate in the study
Arm/Group | Eligible Patients Invited to Participate in the Study
Number analyzed (Participants) | 120
Participants
  Patients that agree to participate | 90
  Patients that refused participation | 30

3. Secondary Outcome: Adequate Randomization
Description: Proportion of patients that were randomized and completed the study
Time Frame: initial clinical visit
Measure: Count of Participants; unit: Participants
Groups:
- Adequate Randomization: Proportion of patients that were post randomization exclusion due to identification of exclusion criteria during the visit
Arm/Group | Adequate Randomization
Number analyzed (Participants) | 90
Participants
  Adequate randomization | 86
  Post Randomization exclusion | 4

4. Secondary Outcome: Completeness of Baseline Survey (Patients)
Description: Proportion of patients that completed the baseline survey
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of Baseline Survey (Patients): Proportion of patients that completed the baseline survey
Arm/Group | Completeness of Baseline Survey (Patients)
Number analyzed (Participants) | 86
Participants
  Completed baseline survey | 84
  Did not complete baseline survey | 2

5. Secondary Outcome: Patient Survey (6 Months)
Description: Proportion of patients that completed the 6 month survey
Time Frame: 6 months
Population: From the initial group of 86 patients, 6 were diagnosed with cancer and not eligible for the follow up survey.
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of 6-month Survey (Patients): Proportion of patients that completed the 6-month survey
Arm/Group | Completeness of 6-month Survey (Patients)
Number analyzed (Participants) | 80
Participants
  Completed the survey | 50
  Did not complete the survey | 30

6. Secondary Outcome: Clinician Baseline Survey
Time Frame: baseline
Population: 17 clinicians care for the patients in the study and were asked to complete a baseline survey
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of Baseline Survey (Clinicians): Proportion of clinicians that completed the baseline survey
Arm/Group | Completeness of Baseline Survey (Clinicians)
Number analyzed (Participants) | 17
Participants
  Completed | 17
  Not Completed | 0

7. Secondary Outcome: Knowledge
Description: To assess knowledge transfer related to thyroid nodules, patients completed a 12-item questionnaire with Yes/No and "I don't know" response options, related to thyroid nodule knowledge. Higher score indicate increased number of correct answers.
Time Frame: baseline
Population: 43 patients were included in each arm, completion of survey items related to knowledge were available for 40 patients in the intervention group and 41 patients in the control group.
Measure: Mean (Standard Deviation); unit: correct response
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 40 | 41
correct response | 72.1 (18.1) | 65.0 (22.4)

8. Secondary Outcome: Decisional Conflict
Description: Decisional conflicts reflects degree of conflict with the decision made. This construct was evaluated with a validated questionnaire that includes 16-items, with the total score transformed into a 1-100 scale, with higher scores indicating greater decisional conflict.
Time Frame: baseline
Population: 43 were randomized in each arm in the study, and for 31 in the intervention group items related the decisional conflict scale in the survey were completed and 23 for those in the control group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 23
score on a scale | 10.9 [0.8 to 42.8] | 20.3 [0 to 29.7]

9. Secondary Outcome: OPTION Score
Description: Observing Patient Involvement (OPTION), evaluates the extent to which clinicians engaged patients in decision making, higher levels more engagement, range (0-100)
Time Frame: baseline
Population: 43 patients were randomized in the study, and clinical visit recordings were available for 42 patients in the intervention group and 43 patients in the control group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 42 | 43
score on a scale | 35.4 [31.3 to 38.5] | 27.1 [20.8 to 30.3]

10. Secondary Outcome: Visit Duration
Description: Length of the clinical visit
Time Frame: baseline
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 42 | 43
minutes | 21.5 (9.3) | 22.1 (9.3)

11. Secondary Outcome: Diagnostic Decision
Description: Proportion of patients undergoing thyroid biopsy
Time Frame: baseline
Population: 43 patients were randomized in the study, the outcome of next diagnostic test (undergoing thyroid biopsy) was assessed from clinical chart review which was available for all patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 43 | 43
Participants
  Thyroid Biopsy | 17 | 22
  Other | 26 | 21

12. Secondary Outcome: Fidelity
Description: Fidelity of use of the conversation aid during clinical visit, evaluating using 12 items during review of clinical visit. Higher percentage refers to higher number of items observed.
Time Frame: baseline
Population: as for outcome 9
Measure: Mean (Standard Error); unit: percentage of items of the conversation
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 42 | 43
percentage of items of the conversation | 78.6 (16.5) | 59.6 (17.9)

13. Secondary Outcome: Risk Communication
Description: Proportion of visits in which thyroid cancer risk was communicated evaluated through review of clinical visit, as yes/no outcome.
Time Frame: baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 42 | 43
Participants
  Risk communicated yes | 39 | 38
  Risk communicated no | 3 | 5

14. Secondary Outcome: Satisfaction With the Communication (Patient)
Description: Likert score, lower number more satisfied, 1-7
Time Frame: baseline
Population: 43 patients were randomized in each arm, for all patients in the intervention group items related to satisfaction were completed in the survey and for 41 in the control group these items were completed in the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 43 | 41
units on a scale | 1.3 (0.8) | 1.4 (0.9)

15. Secondary Outcome: Satisfaction With the Visit (Clinician)
Description: Likert score, higher numbers better, 1-5 options
Time Frame: baseline
Population: Clinicians expressed satisfaction with the clinical visit through a survey, that was completed for all patients in the intervention group (43) and (42) in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 43 | 42
units on a scale | 4.5 (0.7) | 4.4 (0.7)

16. Secondary Outcome: Worry About Thyroid Cancer
Description: Worry about thyroid cancer diagnosis assessed through a survey item, including the options Not at all, rarely/a little or somewhat or a lot
Time Frame: baseline
Population: 43 patients were randomized in each arm, survey responses for this outcome were available for 43 participants in the intervention group and 41 participants in the control group.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Participants received care supplemented by the use of a conversation aid during the clinical visit
- Control Group: Participant received routine care not supplemented by the use of a conversation aid during the clinical visit
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 43 | 41
Participants
  Not at all | 14 | 8
  Rarely/ a litte | 16 | 18
  Somewhat or a lot | 13 | 15

17. Secondary Outcome: Distress Due to Thyroid Nodule (6 Months)
Description: Impact of Event Scale evaluates distress with a new medical situation (new thyroid nodule in this case). The scale includes 6 items, with a score range from 0 to 24 points, with higher values indicating more distress.
Time Frame: 6 months
Population: From the initial population of 86 participants (43 in each group), 6 were diagnosed with thyroid cancer and were not eligible for evaluation of outcomes at 6 months of follow up. Leaving 42 eligible patients in the intervention group (1 cancer diagnosis) of which 29 completed the follow up survey and 38 in the control group (5 cancer diagnoses) of which 21 completed the follow up survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: Patients that received care supplemented by the use of a conversation aid during the visit
- Control Group: Patients that received care without the use of a conversation aid during the clinical visit
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 29 | 21
units on a scale | 1.1 (2.1) | 3.0 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected. Due to the nature of the intervention (conversation aid, used during the clinical visit) adverse events were not collected.
Description: Due to the nature of the intervention (conversation aid, used during the clinical visit) adverse events were not collected.
Groups:
- Clinicians: Clinicians enrolled in the study providing care with or without the conversation aid, according to assigned randomization
Arm/Group | Patient Intervention Group | Patient Control Group | Clinicians
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT04463719/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT04463719/ICF_000.pdf